CLINICAL TRIAL: NCT04803526
Title: Validation of Reproductive Autonomy and Contraceptive Autonomy Scales Among Egyptian Women in Assiut
Brief Title: Validation of Reproductive Autonomy and Contraceptive Autonomy Scales Among Egyptian Women
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Abdelmalek Abdallah, administrator at public health department at faculty of medicine, Assiut university, Assiut University
Other Study IDs: validation study
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to:

1. To validate Arabic version of the reproductive autonomy scale among married women in reproductive age group (15-49 year) in Assiut.
2. To validate Arabic version of the contraceptive autonomy scale among married women in reproductive age group in Assiut

DETAILED DESCRIPTION:
In October 2011, the global population was estimated to be 7 billion. With a growth rate 1.05% per year, the world's population is expected to increase by 2 billion persons in the next 30 years, from 7.7 billion currently to 9.7 billion in 2050 and could peak at nearly 11 billion around 2100 (1). Nearly all of this growth is occurring in developing nations, where fertility rates remain relatively high(2) .

There is an inverse relationship between contraceptive use and fertility. Countries with high proportions of women using contraception generally have lower levels of fertility (3). Globally, 62 percent of married women ages 15 to 49 use a method of family planning and 56 percent use a modern method. These rates are twice as high among women living in high-income countries (67 percent and 60 percent, respectively) compared to women living in low-income countries (34 percent and 29 percent, respectively)(4).

Currently, many more women of reproductive age are using some form of contraception than in 1990. The growing use of contraceptive methods in recent decades has resulted not only in improvements in health-related outcomes such as reduced unintended pregnancies, high-risk pregnancies, maternal mortality, and infant mortality, but also in improvements in schooling and economic outcomes, especially for girls and women. Beyond the impacts of contraceptive use at the individual level, there are benefits at the population level. From a macroeconomic perspective, reductions in fertility enhance economic growth as a result of reduced youth dependency and an increased number of women participating in paid labour(3).

In recognition of the 25th anniversary of the International Conference on Population and Development (ICPD) in 1994, governments reaffirmed the importance of the Program of Action and its further implementation for achieving the Sustainable Development Goals (SDG). The emphasis on universal access to a full range of safe and reliable family planning methods, which help couples and individuals to realize their right to decide freely and responsibly on the number, spacing and timing of births, remains as critical today as it did in 1994(3).

The primary outcome of interest to the family planning community has been contraceptive use (often modern method use), which has traditionally been measured and interpreted in a fairly straightforward way. Generally, a person using a (modern) method is considered a positive outcome, while someone not using a (modern) method is considered a negative outcome (5). Most studies of individual determinants of contraceptive use focus on cognitive, demographic, and contextual variables. However, these models assume that individuals have personal control over their contraceptive behavior(6) .As with other sexual risk outcomes, a woman's capacity to act upon her intention to use contraception may be contingent upon the wishes and actions of her partner or other members of her family or community(7).

Autonomy is defined as the ability of subject to make his/her own decisions without being controlled by anyone else (8). Reproductive autonomy means the women has the power to decide when, if at all, to have children; also, many-but not all-of the choices relevant to reproduction. It means focusing on decisions about whether and when to have children. Women should also generally determine how their pregnancy will be carried out and how the birth will happen(9).

Reproductive autonomy is central to women's welfare both because childbearing takes place in women's bodies and because they are generally expected to take primary responsibility for child rearing(9). It is one of the main reproductive rights. Unfortunately, such autonomy is a low priority for most societies, or is anathema to their belief systems altogether. This situation is doubly sad because women's reproductive autonomy is intrinsically valuable for women and also instrumentally valuable for the welfare of humankind(9).

Recent American study has developed and validated an English multidimensional quantitative instrument that can measure reproductive autonomy. Fourteen items were selected through factor analysis and grouped into three subscales under the construct of reproductive autonomy, labeled "freedom from coercion,""communication," and " decision-making". The scale is considered a reliable instrument to assess a woman's power to control matters regarding contraceptive use, pregnancy, and childbearing, and to evaluate interventions to increase women's autonomy domestically and globally(6).

Reproductive autonomy cannot exist without attention to context to supports, to barriers, to social policy, to social norms(10).

A cross-sectional study of reproductive-age, sexually active women was conducted in Vietnam. It aimed to validate the Reproductive Autonomy Scale among Vietnamese females. Subscales had moderate to high internal consistency (Cronbach's alpha: decision-making power 0.65, freedom from coercion 0.85, and communication ability 0.87). However, the study highlight the need to develop and validate a new measure for reproductive autonomy for populations outside the United States or to adapt the existing measure for these contexts(7).

Although countless approaches to measuring the success of family planning programs exist and novel measures are being continuously introduced, the most widely measured indicators in global family planning continue to be: 1) the total fertility rate; 2) the contraceptive prevalence rate; and 3) unmet need for contraception. These three population-based indicators have the advantage of being routinely measured within nationally representative surveys such as the Demographic and Health Surveys (DHS) around the world without the need for a dedicated study in any given context. In the absence of more nuanced data, we routinely summarize TFR, CPR, and unmet need to paint a picture of the overall family planning context. However, none of these indicators is a measure of health, quality, access, or rights(5).

Clinicians and others show respect to autonomous persons by giving "weight to their considered opinions and choices" and by "refraining from obstructing their actions unless they are clearly detrimental to others(10).

A Novel Family Planning Indicator is the contraceptive autonomy. It is defined as factors necessary for a person to decide for themself what they want in relation to contraception and then to realize that decision, this indicator divides the contraceptive autonomy construct into subdomains of informed choice, full choice and free choice. It aimed to promote reproductive health and right. By acknowledging that autonomous nonuse is a positive outcome, aiming to maximize contraceptive autonomy rather than use could help shift incentives for family planning programs and reduce some common forms of contraceptive coercion, as this measurement approach is realigned with a focus on high-quality rights-based care (6).

Improvements in the status and empowerment of women is central to progress in global development efforts and, perhaps more importantly, to the achievement of equitable treatment and representation of the 3.5 billion women in the world (11). Women's autonomy is an important determinant of women's health and well-being, (12). Review of literature reported the positive associations between women's empowerment and modern contraceptive use and access to maternal interventions such as antenatal care and skilled birth attendance(13), lower fertility, longer birth intervals, and lower rates of unintended pregnancy (11).

Analysis of Pakistani Reproductive Health and Family Planning Survey, 2000 which interviewed a national sample of ever married women aged 15-49 years showed that decision autonomy was significantly associated with both lifetime and current contraception use. On other hand, movement autonomy was not consistently associated with contraceptive use(14).

Omani study analyzed the correlates of women's empowerment and the effect of empowerment on unmet need for contraception. Two indicators of empowerment were used: women's involvement in decision-making and freedom of movement. The results reveled that empowered women were more likely to use contraception(15).

Egypt situation In 2021, the estimated Egypt total population is 101,6 million.(16) Between 2011 and 2018, 11 million people were added to the Egyptian population.(17) Unless the fertility rate of 3.47 changes, by 2030, Egypt's population is expected to grow to 128 million.(18) High fertility contributes to rapid population growth, which threatens the health and well-being of the Egyptian people. In addition, It is likely to impose a costly burden for Egypt by hindering economic development, limiting access to education, food, employment, and potable water, and increasing health risks for women and children.(19) EDHS 2014 findings revealed that 58.5 percent of currently married women in Egypt are currently using a contraceptive method and in Upper Egypt was 50%, modern methods 56.9%, traditional methods 1.6%, total unmet need 12.6%, and not using 41.5%.(20) Women's autonomy over time is a product not only of their individual characteristics, but also of the household and community environment in which they live. Secondary analysis study used the 2006 and 2012 Egyptian Labor Market Panel Survey (ELMPS) and multilevel models. It showed that There are large and consistent variations in women's autonomy by household region of residence and wealth. women in the rural and urban Upper Egypt region are less autonomous than women in the Cairo region, and women in wealthier households are less autonomous compared to the poorest households.(12) The ELMPS measures of autonomy include a set of questions on: (a) participation in household decision-making, (b) woman's ability to move around on her own (mobility), and (c) access to financial resources. (12) Attitudinal measures like attitudes towards gender norms and tolerance of Intimate partner violence are also commonly used as measures of women's empowerment globally(21) A secondary analysis of EDHS 2008 data aimed to assess women's autonomy on modern contraceptive use and its associated factors among Egyptian women. The study revealed that women's autonomy influences their use of modern contraception methods, where household decision-making autonomy was significantly associated with current modern contraceptive use. Women with intermediate and high autonomy were 1.19 (95%CI 1.04-1.35) and 1.32 (95% CI 1.18-1.49) more likely to use modern contraception methods compared to women with low autonomy.(22)

ELIGIBILITY:
Inclusion Criteria:

* Currently married women within reproductive age group (15-49 years)

Exclusion Criteria:

* Current pregnant women, breast feed women (till 6 months), intension to get pregnant within the next 12 months and husband is traveler.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Currently married women within reproductive age group (15-49 years) coming for immunization of their children.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
measuring the internal consistency of the two autonomy scales( reproductive - contraceptive) | 1 year
  by using the cronbach,s alpha

REFERENCES:
- [Background] Nguyen N, Londeree J, Nguyen LH, Tran DH, Gallo MF. Reproductive autonomy and contraceptive use among women in Hanoi, Vietnam. Contracept X. 2019;1:100011. doi: 10.1016/j.conx.2019.100011. PMID 32494775
- [Background] Upadhyay UD, Dworkin SL, Weitz TA, Foster DG. Development and validation of a reproductive autonomy scale. Stud Fam Plann. 2014 Mar;45(1):19-41. doi: 10.1111/j.1728-4465.2014.00374.x. PMID 24615573